CLINICAL TRIAL: NCT04292379
Title: An Innovative Model of Pediatric Acute Mental Health and Addictions Care to Increase Value to Children,Youth, and the Healthcare System
Brief Title: An Innovative Model of Pediatric Acute Mental Health and Addictions Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00092862; REB19-0357 (Other: University of Calgary)
Record Dates: First submitted 2020-02-27; First posted 2020-03-03 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Mental Health; Mental Disorders; Pediatrics; Emergency Psychiatric
Keywords: Emergency Psychiatric Services; Healthcare Delivery
MeSH Terms: conditions — Psychological Well-Being; Mental Disorders | interventions — Standard of Care; Patient Care Bundles

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental study design conducted in three phases. Phase 1 involves standard care. Phase 2 involves introducing a new care bundle to clinical practice using quality improvement and change management strategies. Phase 3 involves delivery of the care bundle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Active Comparator): Mental health visits involve an assessment by a triage nurse who classifies visit urgency into one of five acuity levels using the Canadian Triage and Acuity Scale (CTAS) score. Following triage, children could be assessed by a range of health care providers: emergency department nurse, emergency department physician, mental health nurse, and/or a child and adolescent psychiatrist. Standardized tools are not typically used to guide assessments. Most discharge instructions require families to organize the child's follow-up care.
  Interventions: Other: Standard care
- Care Bundle (Experimental): The bundle standardized suicide risk screening at triage, introduced a focused mental health assessment to guide discussions across health care providers, and included a booked follow-up appointment after the emergency department visit.
  Interventions: Other: Care Bundle

INTERVENTIONS:
Other: Standard care — Standard procedures and assessments
  Arms: Standard care
Other: Care Bundle — Suicide risk screening tool, mental health assessment tool, follow-up appointment
  Arms: Care Bundle

SUMMARY:
The investigators will implement and evaluate an integrated, evidence-based bundle of family-centred, pediatric emergency mental health and addictions care.

DETAILED DESCRIPTION:
The investigators will implement and evaluate an integrated, evidence-based bundle of family-centred, emergency mental health and addictions care. This care bundle will provide high value to families, matching resources and services to need while eliminating healthcare inefficiencies and closing care gaps. The bundle will introduce two well-established tools for healthcare providers to use in EDs, walk-in clinics, and urgent mental health care appointments. These tools are the Ask Suicide-Screening Questions (ASQ) and HEADS-ED, an assessment mnemonic (Home; Education & Employment; Activities & Peers; Drugs & Alcohol; Suicidality; Emotions & Behaviours; Discharge or Current Resources).

The bundle will also introduce new processes to improve healthcare system efficiencies, navigation and transitions between healthcare sectors. For families who receive care in the ED, the investigators will remove the physician gatekeeper role so that children/youth who are screened as low-risk will be offered a follow-up appointment in an urgent mental health care clinic within 24-48 hours. Those who screen as high-risk will see a mental health specialist and undergo a HEADS-ED assessment. Families who follow up in the clinic will receive care that applies a Choice And Partnership Approach (CAPA). CAPA is a collaborative approach to healthcare, where healthcare providers work in partnership with children/youth and their parents to identify choices for care that best match individual needs and preferences.

Study Goal: The investigators' goal is the right care, with the right people, at the right place and time.

Study Design: To measure the bundle's impact, the investigators will use an interrupted time series (ITS) design.

ELIGIBILITY:
Inclusion Criteria:

* Patient is under 18 years of age
* Patient came to the emergency department with a mental health and/or addiction concern
* Patient presented with one of the following CEDIS complaints:

Anxiety, bizarre behaviour, concern for patient's welfare, deliberate self-harm, depression/suicidal, homicidal behaviour, insomnia, pediatric disruptive behaviour, situational crisis, violent behaviour

Exclusion Criteria:

* Brought to the ED by police, peace officer or EMS?
* Held under Form 10
* Features of schizophrenia, schizotypal and delusional disorders (e.g., hallucinations, delusions, active psychosis)
* Behavioural syndromes or other medical concerns requiring medical clearance (e.g., eating disorders)
* Significant self-harm requiring medical clearance (e.g., deep laceration, ingestion, hanging)
* Barriers to communication at triage (e.g., language)
* Previous participation in the study

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1992 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Patient wellbeing at 30 days | 30 days after the index emergency department (ED) visit
  Measured in survey completed by the participant using the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) for patients ≥14 years of age, and the Stirling Children's Wellbeing Scale (SCWBS) for patients <14 years of age.
  For the WEMWBS, each item is scored on a range from 1 to 5. The resulting total score will be between 14 and 70, with lower scores indicating poor wellbeing, and higher scores indicating greater wellbeing. Very low wellbeing is defined as a score of ≤ 45. A substantial decrease in wellbeing is defined as a decrease by 5 or more points.
  For the SCWBS, each item is scored on a range from 1 to 5. The resulting total score will be between 12 and 60, with lower scores indicating poor wellbeing, and higher scores indicating greater wellbeing. Very low wellbeing is defined as a score of ≤ 30. A substantial decrease in wellbeing is defined as a decrease by 5 or more points.

SECONDARY OUTCOMES:
Patient wellbeing at 90 and 180 days | 90 days, and 180 days after the index ED visit
  Measured in survey completed by the participant using the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) for patients ≥14 years of age, and the Stirling Children's Wellbeing Scale (SCWBS) for patients <14 years of age.
  For the WEMWBS, each item is scored on a range from 1 to 5. The resulting total score will be between 14 and 70, with lower scores indicating poor wellbeing, and higher scores indicating greater wellbeing. Very low wellbeing is defined as a score of ≤ 45. A substantial decrease in wellbeing is defined as a decrease by 5 or more points.
  For the SCWBS, each item is scored on a range from 1 to 5. The resulting total score will be between 12 and 60, with lower scores indicating poor wellbeing, and higher scores indicating greater wellbeing. Very low wellbeing is defined as a score of ≤ 30. A substantial decrease in wellbeing is defined as a decrease by 5 or more points.
Family functioning | 30 days after the index ED visit
  Measured in survey completed by the participant using the Family Quality of Life Scale (FQOL). The 25-item scale uses a 5-point rating with a maximum score of 125 indicating highest quality of life.
Satisfaction with acute mental health and addictions ED care | 72 hours after the index ED visit
  Measured in survey completed by the participant using the Service Satisfaction Scale 10 (SSS-10). The scale consists of 12 items (parent version) or 10 items (youth version). Items are scored on a 5-point response scale with a total possible score of 60 (parent) or 50 (youth). Higher scores indicate higher satisfaction.
Proportion of children/youth admitted to child mental health service (child and adolescent psychiatry, mental health team, etc.) | Index ED visit (Day 0)
  Measured using data collected in the patient electronic medical record
Length of ED stay for discharged patients with any mental health presenting complaint | Hours spent in the ED, measured at the index ED visit (Day 0)
  Measured using data collected in the patient electronic medical record. ED Length of stay is defined as the time between patient triage and discharge from the emergency department
Proportion of ED revisits within 72 hours and 30 days for mental health and substance use disorders | 72 hours and 30 days after the index ED visit (Day 0)
  Measured using data collected in the patient electronic medical record

OTHER OUTCOMES:
Death by suicide within 30 days of the index ED visit | 30 days after the index ED visit
  Measured using coroner's data

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Newton, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Derived] Newton AS, Thull-Freedman J, Xie J, Lightbody T, Woods J, Stang A, Winston K, Larson J, Wright B, Stubbs M, Morrissette M, Freedman SB; Pediatric Emergency Research Canada (PERC). Outcomes Following a Mental Health Care Intervention for Children in the Emergency Department: A Nonrandomized Clinical Trial. JAMA Netw Open. 2025 Feb 3;8(2):e2461972. doi: 10.1001/jamanetworkopen.2024.61972. PMID 40009377
- [Derived] Freedman S, Thull-Freedman J, Lightbody T, Prisnie K, Wright B, Coulombe A, Anderson LM, Stang AS, Mikrogianakis A, VanRiper L, Stubbs M, Newton A; Pediatric Emergency Research Canada (PERC). Introducing an innovative model of acute paediatric mental health and addictions care to paediatric emergency departments: a protocol for a multicentre prospective cohort study. BMJ Open Qual. 2020 Dec;9(4):e001106. doi: 10.1136/bmjoq-2020-001106. PMID 33318032